CLINICAL TRIAL: NCT02031406
Title: Impact of Pharmacist Post-discharge Phone Calls on Hospital Readmission and Patient Medication Literacy and Adherence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial initiated, but data collection was inadequate. Analysis was terminated.
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Josh Pevnick, Assistant Professor, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KL2TR000122-00034358; KL2TR000122 (NIH)
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Medication Adherence & Literacy to Predict Readmission; Post-discharge Pharmacist Counseling to Prevent Readmissions
MeSH Terms: conditions — Medication Adherence

ARMS (2):
- Usual care (No Intervention): No extra post-discharge pharmacist counseling is explicitly provided to patients, although some patients may receive it depending on their care setting
- Post-discharge pharmacist counseling (Experimental): Patients will receive post-discharge telephonic pharmacist counseling at around 72 hours after hospital discharge.
  Interventions: Other: Post-discharge counseling on medication adherence & literacy

INTERVENTIONS:
Other: Post-discharge counseling on medication adherence & literacy
  Arms: Post-discharge pharmacist counseling

SUMMARY:
A significant portion of avoidable healthcare expenditures has been attributed to preventable hospital readmissions; thus, reducing hospital readmission rates has become a national healthcare agenda item. Despite much study of this topic, efforts to date have not been especially fruitful in either predicting which patients will require hospital readmission. Preventing readmissions has been even more difficult.

We recently examined a pharmacist intervention that assessed patients' medication literacy and adherence at hospital admission. In this retrospective data, low medication adherence levels were predictive of hospital readmission. There was a non-significant trend between low medication literacy and increased hospital readmissions.

We have now decided to prospectively study this intervention. Prospective study will allow for several improvements on our prior work.

1. We have consulted the literature to more carefully examine existing instruments to measure medication adherence and literacy. Based on this review, and based on our prior results, we have made adjustments to these instruments which should improve reliability, validity, and granularity.
2. In our retrospective work, our intervention of pharmacist counseling was not randomized. Although there were large differences in readmission rates between the patients selected to receive counseling and those who were not thought to require it, there may have been unmeasured confounding variables. Randomizing this intervention will greatly enhance the likelihood that we are comparing two similar groups of patients.

ELIGIBILITY:
Inclusion Criteria:

≥10 chronic prescription medications On anticoagulants Diagnosis of CHF, AMI On narrow therapeutic index drugs E.g. valproic acid, phenytoin, lithium, digoxin History of transplant AND not admitted by transplant team

Exclusion Criteria:

Trauma patients Pediatric patients History of transplant and admitted to the transplant team Patients admitted from or discharged to a SNF or hospice Non-English speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Readmissions | 30 days

SECONDARY OUTCOMES:
Medication Adherence | 30 days after discharge
  Using the Morisky Medication Adherence Scale
Medication Literacy | 30 days
  Using a novel measure of medication literacy

CONTACTS AND LOCATIONS:
Overall Officials: Josh Pevnick, MD, MSHS, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States